CLINICAL TRIAL: NCT00877071
Title: LC Drug Eluting Bead for Regional Chemoembolization to Downstage Unresectable Hepatocellular Carcinoma (HCC) to Liver Transplantation
Brief Title: LC Drug Eluting Bead for Treatment of Liver Cancer Which Cannot be Surgically Removed
Acronym: HCC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Biocompatibles UK Ltd (Industry)
Responsible Party: Principal Investigator, David Geller, MD, David Geller, PI, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO08070016
Record Dates: First submitted 2009-04-04; First posted 2009-04-07 (Estimated); Results first posted 2016-02-08 (Estimated); Last update posted 2016-03-11 (Estimated); Status verified 2016-02

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- LC Drug Eluting Bead, Regional Chemoembolization (Experimental): Use of LC Drug-Eluting Beads for chemoembolization will provide a method for downstaging patients with hepatocellular carcinoma which is not amenable to surgical resection or local ablative therapy to liver transplant eligibility
  Interventions: Drug: LC Bead loaded with doxorubicin

INTERVENTIONS:
Drug: LC Bead loaded with doxorubicin — LC Bead is a new product specifically designed for TACE. LC Bead microspheres will be loaded with between 50-100mg of doxorubicin for each of several TACE procedures. The bead will utilize embolic induced ischemia as well as local chemotherapy in an effort to downstage unresectable HCC to liver transplantation
  Other Names: LC Bead

SUMMARY:
Advanced HCC represents a high unmet medical need with a poor prognosis and few therapeutic options. Patients who present with HCC beyond the currently accepted Milan criteria are not eligible to be listed for liver transplantation. The proposed study offers local regional therapy to a defined population of patients beyond Milan criteria as an attempt to downstage them to eligibility for liver transplant.

DETAILED DESCRIPTION:
LC BeadTM is a new product specifically designed for TACE. LC BeadTM microspheres can be loaded with doxorubicin (Trade name: adriamycin), a chemotherapeutic anthracycline glycolide agent widely accepted for treatment of HCC. This novel bead slowly releases the ionically bound chemotherapeutic agent rather than administering a bolus of chemotherapy as is the case with many alternative methods of TACE. Thus, the LC BeadTM offers the potential advantage of less toxicity and prolonged tumor exposure.

This study offers local regional therapy to a defined population of patients beyond transplant criteria as an attempt to downstage them to eligibility for liver transplantation. This study will make an important contribution to understanding the beads' local effect as seen in the explanted livers of those patients who go on to receive a liver transplant. Additionally, we will examine the impact of this novel treatment tool on patients' quality of life.

ELIGIBILITY:
* Adults patients (≥ 18 years of age) with a diagnosis of HCC that is not amenable to surgical resection or local ablative therapy
* Histological confirmed HCC or clinical/laboratory diagnosis of HCC or nodules larger than 2cm with typical vascular features or AFP > 200
* Patient must have one lesion < 8cm or up to five lesions with total diameter < 8cm
* Quantifiable disease limited to the liver; 40% of liver must be free of tumor burden
* Patient must have at least one tumor lesion that meets both of the following criteria:

  * Lesion can be accurately measured in at least one dimension according to RECIST criteria
  * Lesion has not been previously treated with surgery, radiation therapy, radiofrequency ablation, percutaneous ethanol or acetic acid injection, or cryoablation.
* ECOG performance status ≤ 2
* No prior systemic chemotherapy
* At least 4 weeks since prior TACE or interferon
* Not pregnant
* No significant baseline liver dysfunction. Child-Pugh class A and B 7-8 (in abscence of ascites)
* No significant renal impairment (creatinine clearance < 30mL/minute) or patients on dialysis
* No current infections requiring antibiotic therapy
* Not on anticoagulation or suffering from a known bleeding disorder
* No unstable coronary artery disease or recent MI
* The following laboratory parameters

  * Hemoglobin ≥ 8.5g/dL
  * Total bilirubin ≤ 3.0mg/dL
  * ALT and AST ≤ 5x upper limit of normal
  * Serum creatinine ≤ 1.5x upper limit of normal
  * INR ≤ 1.5 or a PT/PTT within normal limits
  * Platelet count ≥ 50,000/uL
* Ability to understand the protocol and to agree to and sign a written informed consent document

Exclusion Criteria:

* HCC with gross vascular invasion or extrahepatic disease
* Previous or concurrent cancer that is distinct in primary site or histology from HCC except cervical carcinoma in situ, treated basal-cell carcinoma of the skin, superficial bladder tumors (Ta, Tis & T1), and any cancer curatively treated > 3 years prior to entry is permitted
* Renal failure requiring dialysis
* Child-Pugh B9 or C hepatic impairment
* History of cardiac disease: NYHA class 2 congestive heart failure, active coronary artery disease, cardiac arrhythmias requiring anti-arrhythmic therapy other than beta blockers or digoxin, and uncontrolled hypertension. Myocardial infarction more than 6 months prior to study entry is permitted.
* Active clinically serious infections (> CTCAEv3 grade 2)
* Known history of HIV
* Known central nervous system tumors including metastatic brain disease
* History of organ allograft
* Substance abuse (current), psychological, or social conditions that may interfere with the patient's participation in the study or evaluation of the study results.
* Allergy to the investigational agents or any agent given in association with this trial.
* Pregnant or breast-feeding patients. Both men and women enrolled in this trial must use adequate barrier birth control measures during the course of the trial.
* Uncontrolled hypertension defined as systolic blood pressure > 150mmHg or diastolic blood pressure > 90mmHg
* Thrombolic or embolic events such as a cerebrovascular accident including transient ischemic attacks within the past 6 months
* Pulmonary hemorrhage/bleeding event > CTCAE Grade 2 within 4 weeks of first dose of study drug
* Any other hemorrhage/bleeding event > CTCAE Grade 3 within 4 weeks of first dose of study drug
* Serious non-healing wound, ulcer, or bone fracture
* Any contraindication for doxorubicin administration:

  * serum bilirubin > 3mg/dL
  * WBC < 3000 cells/mm3
  * neutrophil < 1500 cells/mm3
  * cardiac ejection fraction < 50 percent assessed by isotopic ventriculography, echocardiography or MRI
  * MUGA scan < 40% ejection fraction
* Any contraindication for hepatic embolization procedures

Excluded therapies and medications, previous and concomitant:

* Prior use of any systemic anti-cancer chemotherapy for HCC
* Prior use of any systemic investigational agents for HCC
* Major surgery within 6 weeks of start of study drug
* Radiotherapy during study or within 3 weeks prior to start of study drug
* Use of biological response modifiers such as granulocyte colony-stimulating factor (G-CSF)within 3 weeks prio to study entry
* Autologous bone marrow transplant or stem cell rescue within four months of study drug initiation
* Concomitant treatment with rifampin or St. John's wort

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2008-11; Primary Completion 2011-05 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David A Geller, MD, Principal Investigator — University of Pittsburgh Medical Center
Locations (1):
- UPMC Liver Cancer Center, Montefiore 7 South, 3459 Fifth Avenue, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | LC Drug Eluting Bead, Regional Chemoembolization
Started | 2
Completed | 0
Not Completed | 2
Not completed — disease progression | 2

BASELINE CHARACTERISTICS:
Arm/Group | LC Drug Eluting Bead, Regional Chemoembolization
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: The Number of Patients in the Cohort Effectively Downstaged to Transplant Eligibility With the LC BeadTM
Description: Advanced HCC represents a high unmet medical need with a poor prognosis and few therapeutic options. Patients who present with HCC beyond the currently accepted Milan criteria are not eligible to be listed for liver transplantation. The proposed study offers local regional therapy to both a defined population of patients beyond Milan criteria as an attempt to downstage them to eligibility for liver transplant as well as those individuals within Milan criteria as an attempt to maintain their eligibility.
Time Frame: 36 months
Population: The data was not analyzed due to insufficient enrollment. A total of 2 patients were enrolled during the course of the study. Both patients experienced disease progression; one patient following Treatment #1 and the other after Treatment #3.
Arm/Group | LC Drug Eluting Bead, Regional Chemoembolization
Number analyzed (Participants) | 0

2. Secondary Outcome: The Objective Tumor Response Rate in Patients With HCC Treated With LC BeadTM Using EASL and RECIST Criteria
Time Frame: 36 months
Population: as for outcome 1
Arm/Group | LC Drug Eluting Bead, Regional Chemoembolization
Number analyzed (Participants) | 0

3. Secondary Outcome: Symptomatic and Quality-of-life Measures in Patients Treated With the LC BeadTM
Time Frame: 36 months
Population: as for outcome 1
Arm/Group | LC Drug Eluting Bead, Regional Chemoembolization
Number analyzed (Participants) | 0

4. Secondary Outcome: The Local Effects of the LC BeadTM in the Explanted Liver of Those Patients Who go on to Receive Liver Transplantation
Time Frame: 36 months
Population: as for outcome 1
Arm/Group | LC Drug Eluting Bead, Regional Chemoembolization
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | LC Drug Eluting Bead, Regional Chemoembolization
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LC Drug Eluting Bead, Regional Chemoembolization (N=2)
hiccoughs (General disorders) | 1 (1)
constipation (Gastrointestinal disorders) | 1 (1)
rectal bleeding (Gastrointestinal disorders) | 1 (1)
diarrhea (Gastrointestinal disorders) | 1 (1)
fever (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No